CLINICAL TRIAL: NCT06177210
Title: Putting Type 2 Diabetes Into Remission: Developing a Person-centred, Interdisciplinary Nutrition Intervention
Brief Title: Type 2 Diabetes Remission
Status: Active, not recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: University of Manitoba (Other)
Responsible Party: Principal Investigator, Jonathan Little, Dr Jonathan Little, University of British Columbia
Other Study IDs: H22-00478
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes Mellitus Remission
Keywords: type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lifestyle intervention: Participants who achieved type 2 diabetes (T2D) remission through lifestyle interventions.
- Bariatric surgery: Participants who achieved type 2 diabetes (T2D) remission through bariatric surgery.

SUMMARY:
The study aims to establish a cohort of patients with type 2 diabetes (T2D) who have achieved remission through lifestyle intervention or bariatric surgery. Remission is defined as a return of HbA1c to less than 6.5% that occurs spontaneously or following an intervention and in the absence of usual glucose-lowering pharmacotherapy for at least 3 months.

DETAILED DESCRIPTION:
The first aim of the study will be to recruit individuals (initial recruitment N=10-12 per group) with physician diagnosed T2D who have achieved remission (HbA1c less than 6.5% and absence of glucose-lowering pharmacotherapy for at least 3 months) through lifestyle interventions or bariatric surgery.

Participants will be recruited by Dr Oliveira:

* from past trials: from previous Informed consent document with ethics approval, Dr Oliveira will approach participants directly through individual email to advise them that a study is being conducted and to enquire if the participant would like to find out more information concerning it.
* via partner/stakeholder networks - Healthcare professionals (e.g., private physician, dietitian, or pharmacist offices): permission to release the contact information will be obtained from the participant by the healthcare professionals before the researcher can use the information for recruitment purposes. The healthcare professionals will either verbally ask the prospective participants' permission to release their names to the Investigator, or distribute an introductory letter describing the study to the prospective participants, with details on how to contact the Investigator if they are interested in participating.
* online advertising: the recruitment poster as per section 9, will be posted on local online newspapers and by posting Recruitment poster on social media.
* website recruitment: https://diabeticstudy.net/index.htm
* In Manitoba: via a recruitment poster as per section 9 that will be circulated via social media and a Letter of initial contact which will be sent to people who express interest in participating.

Inclusion criteria:

1. Have previously been diagnosed with T2D;
2. Have achieved diabetes remission (HbA1c below 6.5% and no glucose lowering medications for at least 3 months)through lifestyle intervention or Bariatric surgery

Exclusion criteria:

1. Have not been diagnosed with T2D;
2. Have an HbA1c level higher than 6.5%;
3. Are taking any glucose lowering medications;
4. Are ongoing medical treatment for diseases such as cancer, auto-immune or inflammatory disease, liver or kidney disorders;
5. Are unable to follow remote guidance by internet or smartphone;
6. Are unable to read or communicate in English.

If demonstrated interest, participants will receive a copy of the Informed Consent by email for their review. If agreed, exclusion and inclusion criteria will be then assessed by completion of an Eligibility Questionnaire and upon confirmation of eligibility, an Electronic Consent form will be signed. The lead researchers will then ensure that the participants understand the details of the study via phone or Zoom call, while asking for confirmation of remission status based on a recent (within 1 month) laboratory A1c value (which is routinely collected by family physicians as part of T2D care). Participants in BC without a current laboratory A1c value will be suggested to ask for an exam request from their family doctor.

Participants will then answer a package of questionnaires:

1. Health Screening Questionnaire + Remission Survey (Lifestyle intervention or Bariatric surgery)
2. Pittsburgh Sleep Quality Index (PSQI)
3. Godin-Shephard Leisure-Time Physical Activity Questionnaire (GSLTPAQ)
4. EQ-5D-5L - Describe and Value Health
5. Three-Factor Eating Questionnaire
6. Perceived Stress Scale

All questionnaires and forms will be sent by REDCap-UBC links and are designed to capture baseline characteristics related to T2D and lifestyle that could influence (or be influenced by) remission.

The second aim of the study is to determine glucose profiles of participants from both groups through CGM.

Participants will receive a study kit at their homes containing a FreeStyle Libre IQ - Continuous Glucose Monitor (CGM) Reader and Sensor, Diet Record papers, and a pre-paid mail envelope. CGM instructions will be sent with the kit and a Zoom meeting can be scheduled to help participants with self-insertion of the device, which is designed to be inserted by persons living with T2D on their own. After completion of the 14-day use, the CGM sensor and reader will be sent back by mail. CGM will serve to confirm some glucose remission criteria stated by the Consensus Report from American Diabetes Association1: mean daily glucose <7.0 mmol/L and 24-h mean glucose concentrations as an estimated HbA1c (eA1C) or most recently named as a glucose management indicator (GMI) <6.5%. The research team is experienced in CGM data collection and analyses having conducted >10 CGM-based studies in the last 8 years.10,11 Once CGM data are analyzed, the research team with follow-up with a Zoom interview in a subsample (n=4-6) of participants in each remission strategy group (lifestyle vs surgery) at each site (n=24 in total). The semi-structured interview will consist of questions that investigate what were the person-level challenges and solutions toward achieving T2D remission. Participants will self-identify in the original consent form if they are willing to participate in the interview portion and the qualitative participants will be recruited based on the lowest and highest values from the CGM analysis (either mean glucose, time-in-range, or glucose standard deviation) whichever gives the largest distribution, the highest and lowest 2-3 from each group (bariatric surgery vs lifestyle) at each site will constitute the sub-sample.

The third aim of the study will be to combine these data with our team's expertise in dietetics, psychology/behavior change, and healthcare delivery, and develop an intervention that meets the needs of patients and healthcare providers that can be embedded into the healthcare system.

The fourth aim (Annual follow-up) is to contact participants from T2D remission cohort for subsequent follow-up, after 1 year. Only participants who consented for future contact and potential future sub-studies that may be conducted once the cohort is established (as per Informed Consent page 5), will be approached. Participation in follow-up study will not be mandatory. Protocol will be similar to first aim study.

ELIGIBILITY:
Inclusion Criteria:

1. Have previously been diagnosed with T2D;
2. Have achieved diabetes remission (HbA1c below 6.5% and no glucose-lowering medications for at least 3 months) through lifestyle intervention and bariatric surgery.

Exclusion Criteria:

1. Have not been diagnosed with T2D;
2. Have an HbA1c level higher than 6.5%;
3. Are taking any glucose-lowering medications;
4. Are ongoing medical treatment for diseases such as cancer, auto-immune or inflammatory disease, liver or kidney disorders;
5. Are unable to follow remote guidance by internet or smartphone;
6. Are unable to read or communicate in English.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who achieved T2D remission
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Establish a cohort of participants who achieved T2D remission through lifestyle interventions | Baseline and after 1 year.
  Establish a cohort of participants who achieved T2D remission through lifestyle interventions.
Establish a cohort of participants who achieved T2D remission through bariatric surgery | Baseline and after 1 year.
  Establish a cohort of participants who achieved T2D remission through bariatric surgery.

SECONDARY OUTCOMES:
Hemoglobin A1C | Baseline and after 1 year.
  Assessed in laboratory exam to confirm diabetes remission status (defined as a return of HbA1c to less than 6.5% that occurs spontaneously or following an intervention and in the absence of usual glucose-lowering pharmacotherapy for at least 3 months).
Questionnaires -Health Screening Questionnaire | Baseline and after 1 year.
  Health Screening Questionnaire: Participants will be asked to answer questions that include age, gender, medical history, and current health status. Questionnaire is included as attachments and will be sent as link from the RedCap platform.
Questionnaires - Pittsburgh Sleep Quality Index (PSQI) | Baseline and after 1 year.
  Pittsburgh Sleep Quality Index (PSQI): is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. Questionnaire is included as attachments and will be sent as link from the RedCap platform
Questionnaires - Perceived Stress Scale | Baseline and after 1 year.
  Perceived Stress Scale: The Perceived Stress Scale (PSS) is a classic stress assessment instrument. It is a 10-item questionnaire originally developed by Cohen et al. (1983) widely used to assess stress levels in young people and adults aged 12 and above. It evaluates the degree to which an individual has perceived life as unpredictable, uncontrollable and overloading over the previous month.
Questionnaires - Godin-Shephard Leisure-Time Physical Activity Questionnaire (GSLTPAQ) | Baseline and after 1 year.
  Godin-Shephard Leisure-Time Physical Activity Questionnaire (GSLTPAQ): allows the assessment of self---reported leisure---time physical activity. The individual is asked to complete a self-explanatory, brief four-item query of usual leisure-time exercise habits. The leisure---time physical activity score is expressed in units and can be computed in two steps. First, weekly frequencies of strenuous, moderate, and mild activities are multiplied by nine, five, and three, respectively; these three latter values correspond to MET (metabolic equivalents) value categories of the activities listed. Then, the total weekly leisure activity score is computed in arbitrary units by summing the products of the separate components.Questionnaire is included as attachments and will be sent as link from the RedCap platform.
Questionnaires - EQ-5D-5L | Baseline and after 1 year.
  EQ-5D-5L: The EQ-5D family of instruments has been developed to describe and value health across a wide range of disease areas. Each EQ-5D instrument comprises a short descriptive system questionnaire and a visual analogue scale (EQ VAS) that are cognitively undemanding, taking only a few minutes to complete. The questionnaire provides a simple descriptive profile of a respondent's health state. Questionnaire is included as attachments and will be sent as link from the RedCap platform.
Questionnaires - Three-Factor Eating Questionnaire (TFEQ) | Baseline and after 1 year.
  Three-Factor Eating Questionnaire (TFEQ): is a self-assessment scale used widely in studies of eating behavior in overweight and normal weight individuals. It was designed to assess three cognitive and behavioral domains (or 'factors') of eating: cognitive restraint (CR), disinhibition and hunger. Questionnaire is included as attachments and will be sent as link from the RedCap platform.
Questionnaires - Remission survey (Bariatric surgery) | Baseline and after 1 year.
  Participants will be asked to answer questions about factors related to putting their type 2 diabetes in remission (different questionnaires for lifestyle intervention and Bariatric surgery).
Questionnaires - Remission survey (Lifestyle intervention) | Baseline and after 1 year.
  Participants will be asked to answer questions about factors related to putting their type 2 diabetes in remission (different questionnaires for lifestyle intervention and Bariatric surgery).
Mean Sensor glucose | Baseline and after 1 year.
  Assessed by continuous glucose monitoring (CGM) device (Abbot FreeStyle Libre IQ) will be inserted by participants into the subcutaneous adipose tissue of the upper arm to collect continuous glucose readings during 14 days.
Minimum sensor glucose | Baseline and after 1 year.
  Assessed by continuous glucose monitoring (CGM) device (Abbot FreeStyle Libre IQ) will be inserted by participants into the subcutaneous adipose tissue of the upper arm to collect continuous glucose readings during 14 days.
Maximum sensor glucose | Baseline and after 1 year.
  Assessed by continuous glucose monitoring (CGM) device (Abbot FreeStyle Libre IQ) will be inserted by participants into the subcutaneous adipose tissue of the upper arm to collect continuous glucose readings during 14 days.
Day time average glucose | Baseline and after 1 year.
  Assessed by continuous glucose monitoring (CGM) device (Abbot FreeStyle Libre IQ) will be inserted by participants into the subcutaneous adipose tissue of the upper arm to collect continuous glucose readings during 14 days.
Standard Deviation (SD) | Baseline and after 1 year.
  Assessed by continuous glucose monitoring (CGM) device (Abbot FreeStyle Libre IQ) will be inserted by participants into the subcutaneous adipose tissue of the upper arm to collect continuous glucose readings during 14 days.
Coefficient of variation (CV) | Baseline and after 1 year.
  Assessed by continuous glucose monitoring (CGM) device (Abbot FreeStyle Libre IQ) will be inserted by participants into the subcutaneous adipose tissue of the upper arm to collect continuous glucose readings during 14 days.
Glucose Management Indicator (GMI) | Baseline and after 1 year.
  Assessed by continuous glucose monitoring (CGM) device (Abbot FreeStyle Libre IQ) will be inserted by participants into the subcutaneous adipose tissue of the upper arm to collect continuous glucose readings during 14 days.
Qualitative interviews | Baseline and after 1 year.
  On a sub-sample of 24 participants, an interview guide adapted from previous studies. It will be followed through a recorded Zoom video call. The main objective is to gather more detailed information regarding participants' process in achieving T2D remission.
  The areas to be investigated will be:
  1. the participant´s experiences and thoughts about their diagnosis and remission;
  2. the information and support given by the health care system and healthcare professionals;
  3. how to manage risks, complications and possible relapse of the disease;
  4. monitoring of glucose levels and other T2D related markers and
  5. lifestyle changes such as diet and exercise. Zoom will be used for video call with participants selected for an interview.

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided